CLINICAL TRIAL: NCT01551654
Title: Non-invasive Acu-point Stimulation (Acu-TENS) in Reduction of Discomfort Associated With Barostat-induced Rectal Distension - a Randomized Controlled Study
Brief Title: Electrical Stimulation Over Acupuncture Points in Reduction of Rectal Discomfort Distension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Wing-Wa Leung, MSc, Mr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRE-2008.546-T
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Pain
Keywords: Pain; Colonoscopy; TENS; Acupuncture
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Acu-TENS (Placebo Comparator): No Electrical output was coming out from the TENS unit
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (ITO Company )
- TENS over acupuncture points (Experimental): A constant mode of electrical stimulation at 2 pulses per second and pulse width at 200µs for 45 minutes. Intensity was set to just initiate muscle contraction.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (ITO Company )

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (ITO Company ) — A mobile small machine for nerve stimulation
  Other Names: (Model 120Z, ITO Company Limited, Tokyo, Japan)

SUMMARY:
Colonoscopy is a stressful and unpleasant procedure especially during the passage of the endoscope through angulations of colon. Electro-acupuncture is one of the alternative to reduce colorectal discomfort. However acupuncture is invasive. This present study explored the effectiveness of a non-invasive treatment modality, Transcutaneous Electrical Nerve Stimulation over Acupuncture points in reduction of colorectal discomfort during barostat-induced rectal distension.

DETAILED DESCRIPTION:
Early colonoscopy screening is encouraged in prevention of development of colorectal cancer as the colonoscopy procedure allows removal of pathological polyps and reduces the risk of cancerous development. While colonoscopy is regarded a minimally invasive procedure, the procedure itself is often associated with abdominal pain and discomfort, especially when the colonoscope is passed through a colonic angulation. The unpleasant feeling during colonoscopy may affect the patient's overall tolerance to the procedure and thereby jeopardizing the accuracy of outcome findings. A combination of narcotic analgesia and benzodiazepines is often used to decrease the abdominal pain and colorectal discomfort during colonoscopy. However these medications are also associated with side effects such as nausea and vomiting. Although uncommon, respiratory and cardiac arrests during colonoscopy were reported. Colonoscopy is now an outpatient day-procedure, unwanted side effects however could prolong recovery time and increase demands of post-intervention nursing care, thereby affecting the cost-effectiveness of the medical model. Undesirable pharmacological side effects have recently led to exploration of alternative management strategies to minimize patient discomfort during colonoscopy.

Electroacupuncture (EA) is widely accepted in China and is considered worldwide a possible treatment option for acute and chronic pain of various origins. The role of acupuncture in managing pain and anxiety during colonoscopy however is unclear. A randomized sham-controlled study (involving 30 patients) suggested that patients receiving EA to acupoints including Zusanli (stomach meridian ST-36) and Hegu (large intestine meridian LI-4) had lower pain level during colonoscopy than those receiving sham acupuncture (SA), but the difference was non-significant statistically. Recently the investigators have shown that application of 45 minutes of EA to Hegu (LI4), Neiguan (PC6) and Zusanli (ST36) was able to effectively reduce colorectal discomfort during Barostat-induced rectal distension. Acupuncture however is invasive, and its application requires an experienced acupuncturist.

Application of Transcutaneous electrical nerve stimulation (TENS) over acupuncture points (Acu-TENS) is a non-invasive modality and a novel analgesic therapy that combines the advantages of acupuncture and TENS in management of painful conditions. Acu-TENS has been shown to be more effective in reducing postoperative analgesic requirement when compared with TENS at nonacupoints. It is postulated that TENS possibly modulates the noxious stimulus of pain via the control of the 'pain-gate' or through the release of β-endorphin. The efficacy of Acu-TENS in pain-relief during colonoscopy has not been reported.

This current study aims to investigate the effect of Acu-TENS on barostat-induced rectal discomfort. A dual drive barostat device was used to mimic colonoscopy in order to control for the nature, intensity and duration of isobaric distension.

ELIGIBILITY:
Inclusion Criteria:

1. Ages of 18-65 undergoing elective colonoscopy
2. Patients with American Society of Anaesthesiologists grading I-II
3. Informed consent available

Exclusion Criteria:

1. Previous history of colorectal resection and abdominal surgery
2. Patients with irritable bowel syndrome (Rome II classifications)
3. Previous experiences of colonoscopy
4. American Society of Anaesthesiologists grading III or above
5. Renal impairment
6. Emergency colonoscopy
7. Pregnancy
8. Allergy to acupuncture needles or electrode pads
9. Refuse to enroll into the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Mean Pain Thresholds | 3 minutes
  During each 60-second phase of sustained incremental pressure, the subject was asked to rate their colorectal sensation using an electronic panel attached to a computer during the resting 2 minutes. Ratings were "no perception", "first perception of distension", "urge to defecate", "discomfort or pain" and "extreme pain".

SECONDARY OUTCOMES:
Beta-endorphins level | 0 minutes, 45 minutes, 90 minutes, 120 minutes
  Venous blood (3 mL) was drawn (from a cannula inserted into the cubital vein of each subject under aseptic technique) before the randomization process (0 minute), immediately after the 45 minutes intervention (45 minutes), at a distension pressure of 24mmHg (45 minutes) and at the end of the intervention (120 minutes). The blood samples were transferred to EDTA tubes with a 4 ºC ice box to the biochemistry laboratory and centrifuged for further assayed with ELISA kit.
Visual Analogue Scale for rectal discomfort | 3 minutes
  Each subject was also asked to rate the degree of rectal discomfort using a visual analogue scale (VAS) with a 10cm un-graduated line, with words "no discomfort at all" anchored to "0" end and "discomfort cannot be tolerated" anchored to the number "10".

CONTACTS AND LOCATIONS:
Overall Officials: Wing-Wa LEUNG, MSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China